CLINICAL TRIAL: NCT05625282
Title: Plantar Plate Repair for Treatment of Floating Toe: Must we Associate it to Weil Osteotomy?
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IIBSP-FLO-2020-131
Record Dates: First submitted 2022-11-11; First posted 2022-11-22 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-10

CONDITIONS: Floating Toe

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Active Comparator): Weil osteotomy and plantar plate repair
  Interventions: Procedure: Weil osteotomy; Procedure: Plantar plate repair
- intervention (Experimental): Weil osteotomy alone
  Interventions: Procedure: Weil osteotomy

INTERVENTIONS:
Procedure: Weil osteotomy — Open, oblique, distal osteotomy of the metatarsal bone, with screw fixation.
Procedure: Plantar plate repair — Plantar plate reconstruction at metatarsophalangeal area, using sutures.
  Arms: control

SUMMARY:
The aim of this study is to assess if isolated Weil osteotomy for floating toe grade II or III provides results that are not inferior to those obtained with the Weil osteotomy associated with plantar plate repair.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old, minimum
* ability to understand treatment and recovery
* floating toe

Exclusion Criteria:

* age less than 18 years old at the moment of recruiting
* patients who are not able to understand treatment and recovery
* intraoperative diagnosis of plantar plate injury grade 0, I or IV in Nery's classification
* secondary surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Manchester-Oxford Foot Questionnaire (MOXFQ) score at the end of follow-up | 1 year
  Score obtained at Manchester-Oxford Foot and Ankle Questionnaire (0-100, where higher scores mean a worse outcome) one year after surgery.

SECONDARY OUTCOMES:
age | moment of recruiting
sex | moment of recruiting
side | moment of recruiting
  left or right foot
rate of recurrence | 1 month, 3 months, 6 months, 1 year after surgery
rate of complications | 1 month, 3 months, 6 months, 1 year after surgery
  related to surgery
Score obtained at Manchester-Oxford Foot and Ankle Questionnaire (0-100, where higher scores mean a worse outcome) | 3 months, 6 months after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Spain